CLINICAL TRIAL: NCT02057406
Title: Omega 3 for Comorbid Depression and Heart Failure Treatment
Brief Title: Omega 3 for Treatment of Depression in Patients With Heart Failure
Acronym: OCEAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wei Jiang (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Wei Jiang, Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00043654; R34MH097034-01A1 (NIH)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2:1 EPA/DHA (Active Comparator): 400/200 EPA/DHA fish oil 2 grams
  Interventions: Drug: 2:1 EPA/DHA
- High EPA (Active Comparator): Almost pure EPA 2 grams
  Interventions: Drug: High EPA
- Placebo (Placebo Comparator): Matched placebo corn oil capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2:1 EPA/DHA — 400 Eicosapentaenoic acid/200 docosahexaenoic acid fish oil 2 grams
  Other Names: 400 EPA/200 DHA 2 grams
  Arms: 2:1 EPA/DHA
Drug: High EPA
  Other Names: An almost pure Eicosapentaenoic acid 2 grams
  Arms: High EPA
Other: Placebo
  Other Names: Matched placebo corn oil capsules
  Arms: Placebo

SUMMARY:
Omega 3 supplements will improve depressive symptoms to a greater extent than placebo in heart failure patients with moderate to severe major depressive disorder.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether (Hypothesis 1a) and how (Hypothesis 1b) the two omega 3 supplements will reduce depressive symptoms in heart failure (HF) patients with moderate-to-severe major depressive disorder (MDD).

Hypothesis 1a: Omega 3 supplements will improve depressive symptoms to a greater extent than placebo; Hypothesis 1b: Pure eicosapentaenoic acid (EPA) will be superior to the EPA: docosahexaenoic acid (DHA) 2:1 in depression improvement.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients, age greater than or equal to 21 years
* Diagnosis of Major Depressive Disorder determined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria with a Hamilton Depression Rating Scale Score greater than or equal to 18*
* New York Heart Association Class greater than or equal to II

  * For patients with with left ventricular ejection fraction greater than 40 %, abnormal brain natriuretic peptide and/or previous hospitalization due to heart failure is also required
  * For inpatients, the Hamilton Depression Rating Scale scores need to be remain at 18 or above for two weeks following the discharge

Exclusion Criteria:

* Significant cognitive impairment, indicated as a Mini-Mental State Examination (MMSE) total score of 23 or lower
* History of alcohol or other drug dependence within the past 90 days
* Severe physical disability (visual, sensory, or motor) that may interfere with psychiatric assessment
* History or presence of psychoses, bipolar disorder, and/or severe personality disorders
* Life-threatening comorbidity with the likelihood of 50% mortality in one year
* Active suicidal ideations
* Current use of antipsychotic medications or psychotropic medications except Selective Serotonin Reuptake Inhibitors (SSRIs) and /or benzodiazepine
* Female patients who have a positive pregnancy test or are lactating. If female patients are of childbearing potential, they must use an effective and accepted means of contraception, such as oral contraceptives or a double-barrier method (condom and diaphragm) to protect against pregnancy
* Documented history of hypersensitivity or intolerance to omega 3 products; or use of omega 3 supplement for greater than or equal to 3 months at an equivalent or greater dose of the proposed study
* Treatment with electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) within 90 days*
* Uncorrected hypothyroidism or hyperthyroidism
* Treatment with any investigational agent within 1 month before randomization
* Acute coronary syndrome, i.e., Myocardial Infarction (MI) or unstable angina, revascularization procedure within the preceding month, or planned cardiac surgery within 3 months postrandomization

  * The exclusion of patients who received ECT or TMS within 90 days is adopted from other depression-intervention trials and meant to eliminate confounders. It is believed that the effects of ECT on mood and cognition may last for a couple of months, and duration of TMS effects is poorly known and may be similar to the ECT intervention.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851
- [Derived] Jiang W, Whellan DJ, Adams KF, Babyak MA, Boyle SH, Wilson JL, Patel CB, Rogers JG, Harris WS, O'Connor CM. Long-Chain Omega-3 Fatty Acid Supplements in Depressed Heart Failure Patients: Results of the OCEAN Trial. JACC Heart Fail. 2018 Oct;6(10):833-843. doi: 10.1016/j.jchf.2018.03.011. Epub 2018 Aug 8. PMID 30098961

RESULTS

PARTICIPANT FLOW:
Groups:
- 2:1 EPA/DHA: 400/200 EPA/DHA fish oil 2 grams
  2:1 EPA/DHA: 400 Eicosapentaenoic acid/200 docosahexaenoic acid (DHA) fish oil 2 grams
- High EPA: Almost pure EPA 2 grams
  High EPA
- Placebo: Matched placebo corn oil capsules
  Placebo
Period: Overall Study
Arm/Group | 2:1 EPA/DHA | High EPA | Placebo
Started | 36 | 36 | 36
Completed | 35 | 33 | 32
Not Completed | 1 | 3 | 4
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Patient transportation issues | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2:1 EPA/DHA | High EPA | Placebo | Total
Number analyzed (Participants) | 36 | 36 | 36 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.73 (16.14) | 58.10 (10.16) | 57.91 (11.68) | 57.92 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 23 | 58
  Male | 21 | 16 | 13 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 15 | 20 | 58
  Black | 13 | 19 | 16 | 48
  Other | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 36 | 108
Treatment Site [Count of Participants; unit: Participants]
  Duke Unviersity Medical Center | 12 | 13 | 13 | 38
  Thomas Jefferson University | 12 | 10 | 10 | 32
  University of North Carolina | 12 | 13 | 13 | 38
Hamilton Depression Rating Scale (HDRS) Score [Mean (Standard Deviation); unit: units on a scale] — The range for the Hamilton Depression Rating Scale is 0 to 52 with higher scores indicating a greater severity of depressive symptoms.
  units on a scale | 22.2 (3.78) | 22.67 (4.24) | 23.56 (4.53) | 22.82 (4.19)
Red Blood Cell/Plasma EPA [Mean (Standard Deviation); unit: percentage of total fatty acids] — Red blood cell/plasma EPA levels are expressed as a percent of total identified fatty acids. Population: All blood samples obtained at baseline for the measurement of EPA were used in this analysis.
  percentage of total fatty acids
    number analyzed (Participants) | 36 | 34 | 35 | 105
    (all) | 0.48 (0.2) | 0.51 (0.24) | 0.49 (0.28) | 0.49 (0.24)

OUTCOME MEASURES:

1. Primary Outcome: Endpoint Hamilton Depression Rating Scale (HAMD) Scores Adjusted for Age, Sex, Treatment Site, and Baseline HAMD Scores.
Description: Endpoint HAMD scores are mean values adjusted for age, race, sex, treatment site, and the baseline HAMD value. The range for the HAMD scores is 0 to 52 with higher scores indicating a greater severity of depressive symptoms.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 2:1 EPA/DHA | High EPA | Placebo
Number analyzed (Participants) | 36 | 36 | 36
units on a scale | 15.1 (0.9) | 15.7 (0.9) | 14.9 (0.9)
Statistical Analysis 1: Comparison: 2:1 EPA/DHA vs Placebo; The model used post-treatment HAMD values as the dependent variable and included age, race, sex, treatment site, and the baseline HAMD value as covariates. This analysis was conducted under intention-to-treat (ITT) in which the missing HAMD endpoint values were imputed using 50 imputations; Test type: Superiority — The EPA/DHA arm versus placebo at Week 12; p = 0.74, ANCOVA
Statistical Analysis 2: Comparison: High EPA vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — High EPA group versus placebo group at Week 12; p = 0.45, ANCOVA

2. Primary Outcome: Endpoint Red Blood Cell/Plasma EPA Values Adjusted for Age, Sex, Treatment Site, and Baseline Red Blood Cell/Plasma EPA Values.
Description: Endpoint EPA values are mean values adjusted for age, race, sex, treatment site, and the baseline EPA value. Red blood cell/plasma EPA values are expressed as a percent of total identified fatty acids.
Time Frame: Week 12
Population: The numbers at baseline reflect the total number of patients who provided samples for the assay of omega 3 percentage of total fatty acids.
  The numbers at endpoint reflect the total number of patients included in the intention to treat analysis.
Measure: Mean (Standard Error); unit: percentage of total fatty acids
Arm/Group | 2:1 EPA/DHA | High EPA | Placebo
Number analyzed (Participants) | 36 | 36 | 36
percentage of total fatty acids | 1.52 (0.15) | 1.86 (0.15) | 0.56 (0.15)
Statistical Analysis 1: Comparison: 2:1 EPA/DHA vs High EPA vs Placebo; The model used post-treatment EPA values as the dependent variable and included age, race, sex, treatment site, and the baseline EPA value as covariates. This analyses was conducted under intention-to-treat (ITT) in which the missing EPA endpoint values were imputed using 50 imputations; Test type: Superiority — Active supplements (2:1 EPA/DHA and High EPA combined) versus placebo at Week 12; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: 2:1 EPA/DHA vs High EPA; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — 2:1 EPA/DHA versus High EPA at Week 12; p = 0.12, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were systematically monitored from enrollment, randomization, at the 12 week intervention and up until 30 days after study drug discontinuation. For patients who terminated from the study before the completion of the 12 week active intervention phase, a 30 day follow-up for AEs was ascertained.
Arm/Group | 2:1 EPA/DHA | High EPA | Placebo
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/36 | 1/36
Serious Adverse Events (participants affected / at risk) | 4/36 | 5/36 | 7/36
Other Adverse Events (participants affected / at risk) | 7/36 | 6/36 | 10/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2:1 EPA/DHA (N=36) | High EPA (N=36) | Placebo (N=36)
Hypertensive Urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Heart Failure Exacerbation (Cardiac disorders) | 2 (2) | 3 (4) | 6 (7)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain on Exertion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mild Stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
(Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Specific cause under review
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2:1 EPA/DHA (N=36) | High EPA (N=36) | Placebo (N=36)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Cataract Removal (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza A (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Right Lower Back/Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Heart failure exacerbation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Arm Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar Burst Fracture, With Acute Exacerbation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes